CLINICAL TRIAL: NCT01982032
Title: Edwards SAPIEN-3 Periprosthetic Leakage Evaluation Versus Medtronic CoreValve in Transfemoral Aortic Valve Implantation (ELECT) Trial
Brief Title: Edwards SAPIEN-3 Periprosthetic Leakage Evaluation Versus Medtronic CoreValve in Transfemoral Aortic Valve Implantation
Acronym: ELECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment, study device unavailable ( CoreValve)
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Pieter Stella, Interventional Cardiologist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL43116.041.13
Record Dates: First submitted 2013-08-27; First posted 2013-11-13 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Periprosthetic Aortic Valve Regurgitation After TAVI
Keywords: Periprosthetic aortic valve regurgitation; 3D transesophageal echocardiography; Cardiac MRI
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Edwards SAPIEN bioprosthesis (Active Comparator): Transcatheter aortic valve replacement with an Edwards SAPIEN bioprosthesis
  Interventions: Procedure: Transcatheter aortic valve replacement; Device: Edwards SAPIEN bioprosthesis
- Medtronic CoreValve® system (Active Comparator): Transcatheter aortic valve replacement with the Medtronic CoreValve system
  Interventions: Procedure: Transcatheter aortic valve replacement; Device: Medtronic CoreValve system

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement
Device: Medtronic CoreValve system — Transcatheter aortic valve replacement with the Medtronic CoreValve system
  Arms: Medtronic CoreValve® system
Device: Edwards SAPIEN bioprosthesis — Transcatheter aortic valve replacement with an Edwards SAPIEN bioprosthesis
  Arms: Edwards SAPIEN bioprosthesis

SUMMARY:
Transcatheter aortic valve replacement (TAVR) is a good alternative treatment for patients with severe aortic valve stenosis with similar mid-term success rates as compared to surgery. Periprosthetic aortic regurgitation (PAR) after TAVR remains an important limitation of this technique. Moderate to severe PAR occurs in 15-45% of the cases and it is an independent predictor of mortality after TAVR. Little is known about potential differences in severity of PAR among different types of aortic valve prosthesis. The current randomized study aims to evaluate potential differences between the Edwards SAPIEN bioprosthesis and the Medtronic CoreValve® system with main focus on PAR and additional focus on other clinical and imaging endpoints. Primary objective of this study is to investigate the difference in the severity of PAR, measured with 3-dimensional transesophageal echocardiography (3DTEE), between patients undergoing the implantation of the Edwards SAPIEN bioprosthesis versus patients receiving the Medtronic CoreValve® bioprosthesis. Secondary objectives of this study include: investigating the value of different imaging modalities in evaluating periprosthetic regurgitation after TAVR and studying the difference in clinical endpoints according to VARC-2 definitions and quality of life after TAVR between two available aortic valve prostheses.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, subjects must meet all of the following criteria:

* Patient is ≥18 years of age and diagnosed with severe symptomatic aortic stenosis, judged inoperable or at high surgical risk (EuroSCORE > 15% or other criteria that make surgery high risk by a consensus among cardiologists and cardiac surgeons in the heart team) and deemed eligible for transfemoral-TAVI.
* Aortic annulus diameter ≥ 18 and ≤ 29 mm as assessed with MSCT.
* No contraindications to study requirements such as MRI or TEE.

Exclusion criteria

* Patients unable or unwilling to give informed consent.
* Patients who are excluded from this study because of the size of their aortic annulus diameter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
PAR (expressed as regurgitant volume [ml]) after TAVR, as diagnosed with 3DTEE | Within 5 days after TAVR
  PAR (expressed as regurgitant volume [ml]) after TAVR, as diagnosed with 3DTEE

SECONDARY OUTCOMES:
PAR (expressed as regurgitant volume [ml]) after TAVR, as diagnosed with cardiac magnetic resonance imaging | Within 5 days after TAVR
  PAR (expressed as regurgitant volume [ml]) after TAVR, as diagnosed with cardiac magnetic resonance imaging
PAR (expressed as regurgitant volume [ml]) 6 months after TAVR, as diagnosed with 3DTEE | At 6 months +/- 2 weeks after TAVR
  PAR (expressed as regurgitant volume [ml]) 6 months after TAVR, as diagnosed with 3DTEE
Clinical endpoints according to the VARC-2 | 30 days, 6months, 1 year
  Clinical endpoints according to the VARC-2
Quality of life, presented as scores of the short form 36 item health status survey (SF-36) | 1 year
  Quality of life, presented as scores of the short form 36 item health status survey (SF-36)
Quality of life, according to the Euroqol questionnaire (EQ-5D) | 1 year
  Quality of life, presented as scores of the Euroqol questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Stella, MD, PhD, Principal Investigator — UMC Utrecht; Pierfrancesco Agostoni, MD, PhD, Study Chair — UMC Utrecht; Nynke Kooistra, MD, Study Director — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Kooistra NHM, Abawi M, Voskuil M, Urgel K, Samim M, Nijhoff F, Nathoe HM, Doevendans PAFM, Chamuleau SAJ, Leenders GEH, Leiner T, Abrahams AC, van der Worp HB, Agostoni P, Stella PR. Randomised comparison of a balloon-expandable and self-expandable valve with quantitative assessment of aortic regurgitation using magnetic resonance imaging. Neth Heart J. 2020 May;28(5):253-265. doi: 10.1007/s12471-020-01414-0. PMID 32246266